CLINICAL TRIAL: NCT04167631
Title: Can Vesical Imaging-Reporting And Data System and Apparent Diffusion Coefficient Values (the VI-RADS/ADC) Accurately Predict Non-Muscle Invasive Bladder Cancer
Brief Title: Can VI-RADS/ADC Accurately Stage Bladder Cancer??
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mahmoud Laymon, Principal Investigator, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MANS.VI-RADS
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: MRI Contrast Media Adverse Reaction; Bladder Cancer; Bladder Disease; Bladder Neoplasm; Bladder Urothelial Carcinoma; Bladder Cancer Stage; Diagnoses Disease
Keywords: VI-RADS; Multiparametric MRI; Non-muscle invasive bladder cancer (NMIBC); Muscle invasive bladder cancer (MIBC)
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urinary Bladder Diseases; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multiparametric MRI (Other): Vesical Imaging-Reporting And Data System (VI-RADS) using multi-parametric MRI.
  Interventions: Radiation: Multi-parametric MRI

INTERVENTIONS:
Radiation: Multi-parametric MRI — Vesical Imaging-Reporting And Data System (VI-RADS) for predicting non-muscle invasive bladder cancer (NMIBC) using multi-parametric MRI.
  Other Names: MP-MRI

SUMMARY:
Vesical Imaging-Reporting And Data System (VI-RADS) is proposed for predicting muscle invasive bladder cancer (MIBC) using multi-parametric MRI. However, No validation study on VI-RADS has been reported yet. Apparent diffusion coefficient (ADC) values on diffusion-weighted MRI are reportedly significantly lower in MIBC than those in non-MIBC(NMIBC).

DETAILED DESCRIPTION:
Vesical Imaging-Reporting And Data System (VI-RADS) is proposed for predicting muscle invasive bladder cancer (MIBC) using multi-parametric MRI. However, No validation study on VI-RADS has been reported yet. Apparent diffusion coefficient (ADC) values on diffusion-weighted MRI are reportedly significantly lower in MIBC than those in non-MIBC(NMIBC).

We aim to examine the accuracy of VI-RADS for predicting MIBC in final histopathology specimen. To assess whether incorporating ADC into VI-RADS improves the MIBC predictive accuracy of VI-RADS

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed at the out-patient cystoscopy with papillary or small nodular bladder tumour

Exclusion Criteria:

* fungating lesions
* beyond the scope of enbloc resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Vesical Imaging-Reporting And Data System (VI-RADS) for discriminating muscle invasive bladder cancer (MIBC) from non-muscle invasive bladder cancer (NMIBC) using multi-parametric MRI. | 18 months
  assessed by final histopathology specimen retrieved by enbloc transurethral resection of bladder tumors (ERBT)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mosbah, MD, Study Chair — Mansoura University; Mohammed Aboelghar, MD, Study Director — Mansoura University
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: No